CLINICAL TRIAL: NCT01423825
Title: A Phase 1 Placebo-Controlled Study Extension to HVTN 073 / SAAVI 102, to Evaluate the Safety and Immunogenicity of Novartis Sub C gp140 Vaccine With MF59 Adjuvant, as a Boost Following SAAVI DNA-C2 Vaccine and SAAVI MVA-C Vaccine, in HIV Uninfected Healthy Adult Participants in South Africa and the United States
Brief Title: Evaluating the Safety and Immune Response to an HIV Vaccine Boost Following the Administration of Two HIV Vaccines, in HIV-Uninfected, Healthy Adults (Study Extension to HVTN 073/SAAVI 102)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: HVTN 073E/SAAVI 102; 11824 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 2011-08-24; First posted 2011-08-26 (Estimated); Last update posted 2021-10-14 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections
MeSH Terms: conditions — HIV Infections | interventions — Sodium Chloride

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Sub C gp140/MF59C.1 Vaccine (Experimental): Participants will receive Sub C gp140 vaccine (100 mcg) admixed with MF59C.1 adjuvant administered as one 0.5 mL injection intramuscularly (IM) in either deltoid at baseline and Month 3.
  Interventions: Biological: Sub C gp140 Vaccine; Biological: MF59C.1 Adjuvant
- Sodium chloride for injection (Placebo Comparator): Participants will receive placebo injection administered as 0.5 mL IM in either deltoid at baseline and Month 3.
  Interventions: Other: Sodium chloride

INTERVENTIONS:
Biological: Sub C gp140 Vaccine — 100 mcg of Sub C gp140 vaccine admixed with MF59C.1 adjuvant administered as one 0.5 mL injection intramuscularly (IM) in either deltoid
  Arms: Sub C gp140/MF59C.1 Vaccine
Biological: MF59C.1 Adjuvant — MF59C.1 adjuvant admixed with 100 mcg of Sub C gp140 vaccine administered as one 0.5 mL injection intramuscularly (IM) in either deltoid. MF59C.1 adjuvant contains no biologicals.
  Arms: Sub C gp140/MF59C.1 Vaccine
Other: Sodium chloride — Sodium chloride as 0.5 mL IM injection in either deltoid to act as placebo
  Arms: Sodium chloride for injection

SUMMARY:
This is an extension of the HVTN 073/SAAVI 102 study. This study will evaluate the safety and immune response to an HIV envelope protein vaccine boost in people who have previously received the SAAVI DNA-C2 and SAAVI MVA-C vaccines or placebo in the HVTN 073/SAAVI 102 study.

DETAILED DESCRIPTION:
The HVTN 073/SAAVI 102 study is evaluating the safety of two experimental HIV vaccines-SAAVI DNA-C2 and SAAVI MVA-C-given sequentially as a prime-boost regimen in healthy, HIV-uninfected adults. This is an extension of that study and will enroll people who participated in the HVTN 073/SAAVI 102 study. Previous studies have shown that a protein vaccine boost to an HIV vaccine may improve antibody responses. This study will evaluate the safety and immune response to an HIV envelope protein vaccine-the Sub C gp140 vaccine with MF59 adjuvant-in healthy, HIV-uninfected adults who have previously participated in the HVTN 073/SAAVI 102 study. Study researchers will explore whether the addition of a protein boost vaccine to the SAAVI DNA-C2 and SAAVI MVA-C vaccine regimen improves antibody response.

This study will enroll people who participated in the HVTN 073/SAAVI 102 study,regardless of whether they received vaccine or placebo. Participants will be randomly assigned to receive either the Sub C gp140 vaccine with MF59 adjuvant or a placebo injection during study visits at baseline and Month 3. At the baseline and Month 3 visits, participants will undergo a physical examination, HIV testing and counseling, pregnancy testing for female participants, interviews and questionnaires, risk reduction counseling, and blood collection (at the baseline visit only). They will then receive their assigned vaccine or placebo as one injection in their upper arm. Participants will remain in the clinic for 30 minutes after receiving the vaccination for observation and monitoring. For 3 days after the vaccination, participants will record any side effects in a symptom log and make contact daily with the study site staff.

Additional study visits will occur at Weeks 1 and 2, 1 and 2 weeks after the Month 3 visit, and Months 6 and 9. At these visits, select baseline study procedures will occur. At Month 15, study staff will contact participants for follow-up health monitoring. Participants will then complete any annual health contacts for the original HVTN 073/SAAVI 102 study.

ELIGIBILITY:
Inclusion Criteria:

* Hemoglobin greater than or equal to 11.0 g/dL
* White blood cell (WBC) count greater than 2,500 cells/mm^3
* Platelets greater than or equal to 125,000/mm^3
* Chemistry panel: alanine aminotransferase (ALT), aspartate aminotransferase (AST), and alkaline phosphatase less than 1.25 times the institutional upper limit of normal; creatinine less than or equal to the institutional upper limit of normal
* Normal urine:

  1. Negative urine glucose, and
  2. Negative or trace urine protein, and
  3. Negative or trace urine hemoglobin (if trace hemoglobin is present on dipstick, a microscopic urinalysis within institutional normal range)
* Able and willing to provide informed consent
* Negative HIV-1 and -2 blood test: Participants must have a negative HIV test result as specified by the HVTN Laboratory Program's in-study HIV diagnostic algorithm
* Participants who were born female: negative serum or urine beta human chorionic gonadotropin (beta-HCG) pregnancy test performed on the day of initial study extension vaccination prior to vaccination
* Reproductive status: A participant who was born female must agree to consistently use effective contraception from at least 21 days prior to enrollment through 90 days after the participant's final vaccination, for sexual activity that could lead to pregnancy. More information on this criterion can be found in the protocol.
* Participants who were born female must also agree not to seek pregnancy through alternative methods such as artificial insemination or in vitro fertilization until after the last scheduled protocol visit
* Receipt of scheduled injection at visit 11 in the HVTN 073/SAAVI 102 study

Exclusion Criteria:

* Participant meets criteria for delay or discontinuation of vaccination or termination from the study. More information on this criterion can be found in the protocol.
* Participant has an unresolved AE that is possibly, probably, or definitely related to the study product
* Any medical, psychiatric, or social condition, or occupational or other responsibility that, in the judgment of the investigator, would interfere with, or serve as a contraindication to, protocol adherence, assessment of safety or reactogenicity, or a participant's ability to give informed consent (e.g., a skin condition overlying a potential injection site, which could interfere with reactogenicity assessment)

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2011-08; Primary Completion 2013-07 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Safety data, including signs and symptoms of local and systemic reactogenicity, laboratory measures of safety, adverse events (AEs), and AEs requiring expedited adverse event (EAE) reporting to DAIDS | Measured through Month 15

SECONDARY OUTCOMES:
HIV-1-specific neutralizing and binding antibody assays at 2 weeks following vaccination with Novartis Sub C gp140 with MF59 | Measured at Months 0.5, 3.5 and 9
Neutralizing antibody breadth against heterologous primary isolates | Measured at Months 0.5, 3.5 and 9

CONTACTS AND LOCATIONS:
Overall Officials: Glenda Gray, Study Chair — University of the Witswatersrand
Locations (4):
- United States (2):
  - Brigham and Women's Hospital Vaccine CRS (BWH VCRS), Boston, Massachusetts
  - Fenway Health (FH) CRS, Boston, Massachusetts
- South Africa (2):
  - Soweto HVTN CRS, Johannesburg, Gauteng
  - Emavundleni CRS, Cape Town, Western Cape

REFERENCES:
- [Background] Rerks-Ngarm S, Pitisuttithum P, Nitayaphan S, Kaewkungwal J, Chiu J, Paris R, Premsri N, Namwat C, de Souza M, Adams E, Benenson M, Gurunathan S, Tartaglia J, McNeil JG, Francis DP, Stablein D, Birx DL, Chunsuttiwat S, Khamboonruang C, Thongcharoen P, Robb ML, Michael NL, Kunasol P, Kim JH; MOPH-TAVEG Investigators. Vaccination with ALVAC and AIDSVAX to prevent HIV-1 infection in Thailand. N Engl J Med. 2009 Dec 3;361(23):2209-20. doi: 10.1056/NEJMoa0908492. Epub 2009 Oct 20. PMID 19843557
- [Background] Evans TG, Keefer MC, Weinhold KJ, Wolff M, Montefiori D, Gorse GJ, Graham BS, McElrath MJ, Clements-Mann ML, Mulligan MJ, Fast P, Walker MC, Excler JL, Duliege AM, Tartaglia J. A canarypox vaccine expressing multiple human immunodeficiency virus type 1 genes given alone or with rgp120 elicits broad and durable CD8+ cytotoxic T lymphocyte responses in seronegative volunteers. J Infect Dis. 1999 Aug;180(2):290-8. doi: 10.1086/314895. PMID 10395842
- [Background] Srivastava IK, Kan E, Sun Y, Sharma VA, Cisto J, Burke B, Lian Y, Hilt S, Biron Z, Hartog K, Stamatatos L, Diaz-Avalos R, Cheng RH, Ulmer JB, Barnett SW. Comparative evaluation of trimeric envelope glycoproteins derived from subtype C and B HIV-1 R5 isolates. Virology. 2008 Mar 15;372(2):273-90. doi: 10.1016/j.virol.2007.10.022. Epub 2007 Dec 3. PMID 18061231
- [Derived] Gray GE, Mayer KH, Elizaga ML, Bekker LG, Allen M, Morris L, Montefiori D, De Rosa SC, Sato A, Gu N, Tomaras GD, Tucker T, Barnett SW, Mkhize NN, Shen X, Downing K, Williamson C, Pensiero M, Corey L, Williamson AL. Subtype C gp140 Vaccine Boosts Immune Responses Primed by the South African AIDS Vaccine Initiative DNA-C2 and MVA-C HIV Vaccines after More than a 2-Year Gap. Clin Vaccine Immunol. 2016 Jun 6;23(6):496-506. doi: 10.1128/CVI.00717-15. Print 2016 Jun. PMID 27098021